CLINICAL TRIAL: NCT07336576
Title: Surgery-Oriented Classification and Treatment Strategy for Adult Congenital Biliary Dilation
Brief Title: Treatment Strategy for Adult Congenital Biliary Dilation
Status: Completed | Type: Observational
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Principal Investigator, Shuo Jin, Associate Chief Physician, Beijing Tsinghua Chang Gung Hospital
Other Study IDs: 25534-0-01
Record Dates: First submitted 2025-12-12; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Congenital Biliary Dilation
Keywords: Choledochal Cyst
MeSH Terms: conditions — Choledochal Cyst

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- underwent surgical treatment for CBD between November 2014 and October 2024
  Interventions: Procedure: hepatectomy、liver transplantation、hepaticojejunostomy

INTERVENTIONS:
Procedure: hepatectomy、liver transplantation、hepaticojejunostomy — resection of the diseased bile duct, elimination of secondary lesions, and restoration of biliary-enteric continuity.

SUMMARY:
The management of congenital biliary dilations (CBDs), including choledochal cysts, represents one of the most challenging areas in hepatobiliary surgery due to their potential implications for long-term morbidity and malignant transformation. While CBDs have a relatively low incidence in Western populations (1/150,000-1/100,000), the prevalence is notably higher in Asian countries (1/1,000), making it a significant global health concern. Although complete surgical resection remains the standard of care, the optimal extent of resection and reconstruction strategy, particularly for complex disease patterns, continues to be debated. To address these challenges, the current study proposes a novel surgery-oriented classification system for adult CBD based on the analysis of 234 consecutive cases.

ELIGIBILITY:
Inclusion Criteria ：

1. Age: Adults (≥18 years).
2. Study population: Consecutive patients treated at Beijing Tsinghua Changgung Hospital.
3. Time frame: Underwent surgical treatment between November 2014 and October 2024.
4. Condition/Procedure: Underwent surgical treatment for common bile duct (CBD) diseases.
5. Diagnostic confirmation: Presence, location, and extent of CBD dilatation were diagnosed by preoperative imaging/radiology, and confirmed intraoperatively. Exclusion Criteria ：

1.Secondary biliary dilatation due to proximal obstruction, including intrahepatic and/or extrahepatic bile duct dilatation caused by proximal biliary obstruction, such as:

1. benign stricture,
2. malignant stricture,
3. obstructive stones.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive adult patients who underwent surgical treatment for common bile duct (CBD) diseases between November 2014 and October 2024 at Beijing Tsinghua Changgung Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 234 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
The modified Mayo Clinic score for CBD | Last follow-up time (assessed up to 10 year)
  Patients were stratified into excellent, good, fair, and poor categories based on established criteria

SECONDARY OUTCOMES:
perioperative complications | Perioperative period（Within 3 months after surgery）
  graded according to the Clavien-Dindo classification,23 specific complications assessed using the International Study Group of Liver Surgery (ISGLS) criteria, including posthepatectomy liver dysfunction, bile leakage, and pancreatic leakage24-26
long-term disease-free survival | Last follow-up time (assessed up to 10 year)
  long-term disease-free survival defined as the interval from surgery to the first occurrence of any of the following events: cholangitis episode, bile stone formation, cholangiocarcinoma development, any long-term complications related to biliary surgery, or death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Hepatopancreatobiliary Center, Beijing Tsinghua Changgung Hospital, Key Laboratory of Digital Intelligence Hepatology, Ministry of Education, School of Clinical Medicine, Tsinghua University, Beijing, China, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No